CLINICAL TRIAL: NCT00432679
Title: Clinical Evaluation of Rosiglitazone Maleate (BRL49653C) in Patients With Type 2 Diabetes Mellitus (Combination Therapy With Sulfonyl Urea) - A Placebo-Controlled Double-Blind Study -
Brief Title: A Study Of BRL49653C For The Treatment Of Type 2 Diabetes (Combination Therapy With Sulfonyl Urea) -With Placebo Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVD105248
Record Dates: First submitted 2007-02-06; First posted 2007-02-08 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: rosiglitazone; Avandia; type 2 diabetes mellitus; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- arm 1 (Experimental): study drug
  Interventions: Drug: Rosiglitazone (BRL49653C)

INTERVENTIONS:
Drug: Rosiglitazone (BRL49653C) — study drug

SUMMARY:
This study was designed to compare the efficacy and safety of BRL49653C versus placebo with concomitant use of sulfonyl urea (SU).

ELIGIBILITY:
Inclusion criteria:

* Patients with type 2 diabetes mellitus managed by SU will be candidate for this study. These candidates will be checked up on their clinical laboratory data, and must have adequate blood, liver and kidney function.

Exclusion criteria:

* Patient with serious cardiovascular disease or serious hepatic disease will not be eligible.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2006-05-24 (Actual); Primary Completion 2007-03-28 (Actual); Study Completion 2007-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Japan (3):
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Ōita
- GSK Investigational Site

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: AVD105248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AVD105248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AVD105248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AVD105248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AVD105248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AVD105248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AVD105248 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 19 April 2006 to 28 March 2007, total of 149 participants were randomized at 22 centers in Japan.
Pre-assignment Details: Out of 172 participants given consent to participate in the study, 23 participants were withdrawn from the study before randomization.
Groups:
- Rosiglitazone 4 mg Orally Once Daily: Participants in this arm were randomized to receive rosiglitazone (BRL49653C) 4 milligrams (mg) tablets orally once daily before or after breakfast for 16 weeks. Participants also received either of concomitant medication (sulphonylureas) glibenclamide (1.25 to 5 mg), gliclazide (40 to 80 mg) or glimepiride (1 to 3 mg) per day during study.
- Placebo: Participants in this arm were randomized to receive rosiglitazone placebo tablets orally once daily before or after breakfast for 16 weeks. Participants also received either of concomitant medication (sulphonylureas) glibenclamide (1.25 to 5 mg), gliclazide (40 to 80 mg) or glimepiride (1 to 3 mg) per day during study.
Period: Overall Study
Arm/Group | Rosiglitazone 4 mg Orally Once Daily | Placebo
Started | 74 | 75
Completed | 69 | 72
Not Completed | 5 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Rosiglitazone 4 mg Orally Once Daily: Participants in this arm were randomized to receive rosiglitazone (BRL49653C) 4 mg tablets orally once daily before or after breakfast for 16 weeks. Participants also received either of concomitant medication (sulphonylureas) glibenclamide (1.25 to 5 mg), gliclazide (40 to 80 mg) or glimepiride (1 to 3 mg) per day during study.
- Total: Total of all reporting groups
Arm/Group | Rosiglitazone 4 mg Orally Once Daily | Placebo | Total
Number analyzed (Participants) | 74 | 75 | 149
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.1 (8.81) | 61.6 (9.80) | 60.8 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 55
  Male | 47 | 47 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 74 | 75 | 149
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) After 16 Weeks of Treatment in Rosiglitazone Group and Placebo Group
Description: Baseline value was value on Day 0. Change from Baseline was defined as value at Week 16 minus Baseline value. The full analysis set used which was defined as remaining after participant who infringed on the following events were excluded from the randomized participants, who did not take the investigational drug during or after the treatment period (amount of investigational drug taken was zero tablets) and who were not measured for HbA1c even once as the observation period Baseline value or in the treatment period (after the investigational drug was prescribed), or for whom the above were unavailable (including cases that the above were considered missing measurements due to a defective sample).
Time Frame: Baseline (Day 0) and Week 16
Population: Full analysis set used.
Measure: Mean (Standard Deviation); unit: Percentage of Glycosylated Hemoglobin
Arm/Group | Rosiglitazone 4 mg Orally Once Daily | Placebo
Number analyzed (Participants) | 74 | 75
Percentage of Glycosylated Hemoglobin | -0.62 (0.074) | 0.19 (0.073)
Statistical Analysis 1: Comparison: Rosiglitazone 4 mg Orally Once Daily vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Change from Baseline in HbA1c = Treatment+ Baseline HbA1c+ Gender+ body mass index (BMI); Mean Difference (Net) = -0.81, 95% CI 2-sided [-1.01 to -0.61], Standard Error of Mean 0.102

2. Secondary Outcome: Change From Baseline After 16 Weeks of Treatment in Fasting Plasma Glucose (FPG)
Description: Baseline value was value on Day 0. Change from Baseline was defined as value at Week 16 minus Baseline value.
Time Frame: Baseline (Day 0) and Week 16
Population: Full analysis set used.
Measure: Mean (Standard Deviation); unit: Mg per decilliter
Arm/Group | Rosiglitazone 4 mg Orally Once Daily | Placebo
Number analyzed (Participants) | 74 | 75
Mg per decilliter | -15.9 (28.91) | 6.2 (32.69)
Statistical Analysis 1: Comparison: Rosiglitazone 4 mg Orally Once Daily vs Placebo; Test type: Superiority or Other; p < 0.001, Unpaired t-test; Mean Difference (Net) = -22.1, 95% CI 2-sided [-32.1 to -12.1], Standard Error of Mean 5.06

3. Secondary Outcome: Change From Baseline After 16 Weeks of Treatment in Fasting Insulin
Description: Baseline value was value on Day 0. Change from Baseline was defined as value at Week 16 minus Baseline value.
Time Frame: Baseline (Day 0) and Week 16
Population: Full analysis set used. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microunits per millilliter
Arm/Group | Rosiglitazone 4 mg Orally Once Daily | Placebo
Number analyzed (Participants) | 74 | 73
Microunits per millilliter | -0.479 (3.2699) | -1.197 (6.1434)
Statistical Analysis 1: Comparison: Rosiglitazone 4 mg Orally Once Daily vs Placebo; Test type: Superiority or Other; p = 0.377, Unpaired t-test; Mean Difference (Net) = 0.718, 95% CI 2-sided [-0.883 to 2.319], Standard Error of Mean 0.8102

4. Secondary Outcome: Change From Baseline After 16 Weeks of Treatment in Fasting Proinsulin
Description: Baseline value was value on Day 0. Change from Baseline was defined as value at Week 16 minus Baseline value.
Time Frame: Baseline (Day 0) and Week 16
Population: Full analysis set used. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picomoles per millilliter
Arm/Group | Rosiglitazone 4 mg Orally Once Daily | Placebo
Number analyzed (Participants) | 74 | 73
Picomoles per millilliter | -1.64 (13.630) | 0.40 (11.666)
Statistical Analysis 1: Comparison: Rosiglitazone 4 mg Orally Once Daily vs Placebo; Test type: Superiority or Other; p = 0.330, Unpaired t-test; Mean Difference (Net) = -2.04, 95% CI 2-sided [-6.18 to 2.09], Standard Error of Mean 2.094

5. Secondary Outcome: Change From Baseline After 16 Weeks of Treatment in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: Baseline value was value on Day 0. Change from Baseline was defined as value at Week 16 minus Baseline value.
Time Frame: Baseline (Day 0) and Week 16
Population: Full analysis set used. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: MilliUnit per liter*millimoles per liter
Arm/Group | Rosiglitazone 4 mg Orally Once Daily | Placebo
Number analyzed (Participants) | 74 | 73
MilliUnit per liter*millimoles per liter | -0.496 (1.5562) | -0.486 (3.7556)
Statistical Analysis 1: Comparison: Rosiglitazone 4 mg Orally Once Daily vs Placebo; Test type: Superiority or Other; p = 0.983, Unpaired t-test; Mean Difference (Net) = -0.010, 95% CI 2-sided [-0.945 to 0.925], Standard Error of Mean 0.4730

6. Secondary Outcome: Change From Baseline After 16 Weeks of Treatment in Homeostasis Model Assessment of Beta-cell Function (HOMA-beta)
Description: Baseline value was value on Day 0. Change from Baseline was defined as value at Week 16 minus Baseline value.
Time Frame: Baseline (Day 0) and Week 16
Population: Full analysis set used. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of normal beta cells function
Arm/Group | Rosiglitazone 4 mg Orally Once Daily | Placebo
Number analyzed (Participants) | 74 | 73
Percentage of normal beta cells function | 3.776 (18.7875) | -4.444 (24.0408)
Statistical Analysis 1: Comparison: Rosiglitazone 4 mg Orally Once Daily vs Placebo; Test type: Superiority or Other; p = 0.022, Unpaired t-test; Mean Difference (Net) = 8.220, 95% CI 2-sided [1.191 to 15.248], Standard Error of Mean 3.5560

7. Secondary Outcome: Change From Baseline After 16 Weeks of Treatment in Adiponectin
Description: Baseline value was value on Day 0. Change from Baseline was defined as value at Week 16 minus Baseline value.
Time Frame: Baseline (Day 0) and Week 16
Population: Full analysis set used. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micrograms per millilliter
Arm/Group | Rosiglitazone 4 mg Orally Once Daily | Placebo
Number analyzed (Participants) | 74 | 74
Micrograms per millilliter | 9.19 (7.030) | 0.98 (2.301)
Statistical Analysis 1: Comparison: Rosiglitazone 4 mg Orally Once Daily vs Placebo; Test type: Superiority or Other; p < 0.001, Unpaired t-test; Mean Difference (Net) = 8.21, 95% CI 2-sided [6.52 to 9.91], Standard Error of Mean 0.860

8. Secondary Outcome: Change From Baseline After 16 Weeks of Treatment in Leptin and High Sensitivity C-reactive Protein (Hs-CRP)
Description: Baseline value was value on Day 0. Change from Baseline was defined as value at Week 16 minus Baseline value.
Time Frame: Baseline (Day 0) and Week 16
Population: Full analysis set used. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per millilliter
Arm/Group | Rosiglitazone 4 mg Orally Once Daily | Placebo
Number analyzed (Participants) | 74 | 74
Nanograms per millilliter
  Leptin | 0.59 (2.751) | -0.07 (1.332)
  Hs-CRP | -189.1 (5376.91) | 699.7 (4349.58)
Statistical Analysis 1: Comparison: Rosiglitazone 4 mg Orally Once Daily vs Placebo; Test type: Superiority or Other; p = 0.069, Unpaired t-test; Mean Difference (Net) = 0.65, 95% CI 2-sided [-0.05 to 1.35], Standard Error of Mean 0.355 — Comparison of leptin
Statistical Analysis 2: Comparison: Rosiglitazone 4 mg Orally Once Daily vs Placebo; Test type: Superiority or Other; p = 0.271, Unpaired t-test; Mean Difference (Net) = -888.8, 95% CI 2-sided [-2477.7 to 700.1], Standard Error of Mean 803.96 — Comparison of hs-CRP

9. Secondary Outcome: Percentage of Participants With Changes in HbA1c and FPG Meeting Specified Criteria After 16 Weeks of Treatment
Description: The specified criteria for HbA1c was, if the decrease from the observation period Baseline value meets the following conditions: 1) decrease from the observation period Baseline value is 0.7% or more; 2) fell below 6.5%; 3) satisfied either 1 or 2 noted above. And for FPG was, if the decrease from the observation period Baseline value meets the following conditions: 1) decrease of 30 mg per decilliter or more from the observation period Baseline value; 2) fell below 126 mg per deciliter; 3) satisfied either 1 or 2 noted above.
Time Frame: Up to Week 16
Population: Full analysis set used.
Measure: Number; unit: Percentage of participants
Arm/Group | Rosiglitazone 4 mg Orally Once Daily | Placebo
Number analyzed (Participants) | 74 | 75
Percentage of participants
  HbA1c, decrease by 0.7% | 44.6 | 4.0
  HbA1c, fell below 6.5% | 6.8 | 0.0
  HbA1c, satisfied either 1 or 2 | 44.6 | 4.0
  FPG, decrease of 30 milligrams per decilliter | 31.1 | 8.0
  FPG, fell below 126 milligrams per deciliter | 16.2 | 9.3
  FPG, satisfied either 1 or 2 | 35.1 | 14.7
Statistical Analysis 1: Comparison: Rosiglitazone 4 mg Orally Once Daily vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 40.6, 95% CI 2-sided [27.1 to 54.1] — Comparison of HbA1c, decrease by 0.7%
Statistical Analysis 2: Comparison: Rosiglitazone 4 mg Orally Once Daily vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 6.8, 95% CI 2-sided [-0.3 to 13.8] — Comparison of HbA1c, fell below 6.5%
Statistical Analysis 3: Comparison: Rosiglitazone 4 mg Orally Once Daily vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 40.6, 95% CI 2-sided [27.1 to 54.1] — Comparison of HbA1c, satisfied either 1 or 2
Statistical Analysis 4: Comparison: Rosiglitazone 4 mg Orally Once Daily vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 23.1, 95% CI 2-sided [9.5 to 36.6] — Comparison of FPG, decrease of 30 milligrams per decilliter
Statistical Analysis 5: Comparison: Rosiglitazone 4 mg Orally Once Daily vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 6.9, 95% CI 2-sided [-5.1 to 18.9] — Comparison of FPG, fell below 126 milligrams per deciliter
Statistical Analysis 6: Comparison: Rosiglitazone 4 mg Orally Once Daily vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 20.5, 95% CI 2-sided [5.6 to 35.3] — Comparison of FPG, satisfied either 1 or 2

ADVERSE EVENTS:
Time Frame: All adverse events (AE) and serious adverse events (SAE) were reported during the clinical trial period (from the observation period (Week -4) to the post-trial examination date (up to Week 18 or 2 weeks after the discontinuation).
Description: Full analysis set was used for reporting non-SAE and SAE.
Arm/Group | Rosiglitazone 4 mg Orally Once Daily | Placebo
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/75
Serious Adverse Events (participants affected / at risk) | 1/74 | 1/75
Other Adverse Events (participants affected / at risk) | 61/74 | 53/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosiglitazone 4 mg Orally Once Daily (N=74) | Placebo (N=75)
Liposacromal recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain stem infarction (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosiglitazone 4 mg Orally Once Daily (N=74) | Placebo (N=75)
Blood creatine phosphokinase increased (Investigations) | 9 | 3
Weight increased (Investigations) | 10 | 1
Blood triglyccrides increased (Investigations) | 7 | 1
Blood pressure increased (Investigations) | 2 | 4
Brain natriuretic peptide increased (Investigations) | 3 | 2
Blood cholesterol increased (Investigations) | 2 | 1
Urine ketone body present (Investigations) | 0 | 3
Blood urine present (Investigations) | 2 | 0
Hjgh density lipoprotein decreased (Investigations) | 2 | 0
Low density lipoprotein increased (Investigations) | 1 | 1
Protein urine present (Investigations) | 0 | 2
Blood albumin decreased (Investigations) | 1 | 0
Blood uric acid increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Monocyte count increased (Investigations) | 1 | 0
Neutrophll count decreased (Investigations) | 1 | 0
Reticulocyte count increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 10 | 12
Pharyngitis (Infections and infestations) | 3 | 3
Cystitis (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Hordeolum (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchitis acute (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Impetigo (Infections and infestations) | 0 | 1
lnfluenza (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Gastritis (Gastrointestinal disorders) | 3 | 0
Reflux ocsophagitis (Gastrointestinal disorders) | 1 | 2
Stomach discomfort (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 1
Periodontitis (Gastrointestinal disorders) | 2 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Duodenal scarring (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 8 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngolaryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Myajgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Oedema peripheral (General disorders) | 6 | 0
Pyrexia (General disorders) | 0 | 2
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Feeling abnonnal (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 3
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0
Tooth injury (Injury, poisoning and procedural complications) | 0 | 1
Thennal bum (Injury, poisoning and procedural complications) | 0 | 1
Neck injury (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Headache (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 2 | 0
Hypoaesthcsia (Nervous system disorders) | 2 | 0
Areflexia (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 2
Cataract (Eye disorders) | 1 | 1
Corneal epithelium disorder (Eye disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Punctate keratitis (Eye disorders) | 0 | 1
Corneal exfoliation (Eye disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0
Bundle branch block right (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Hyperaemia (Vascular disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1
Adrenal mass (Endocrine disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.